CLINICAL TRIAL: NCT02530580
Title: A Phase I Single Site, Single Dose, Randomized, Double-blind, Placebo Controlled, 2-way Cross-over Biomarker Study Investigating the Effect of the GABA Modulator AZD7325 on Cutaneous Sensation in Healthy Volunteers
Brief Title: Effects of GABA Modulator AZD7325 on Cutaneous Sensation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13/0261; 2015-000642-35 (EudraCT Number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-21 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: GABA modulator; AZD7325; Object manipulation; Cutaneous sensation; Manual dexterity
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 mg AZD7325 (Experimental): 10 mg AZD7325 in orange capsule, Size 0, 2 capsules as a single oral dose
  Interventions: Drug: 20 mg AZD7325; Drug: Placebo
- Placebo (Placebo Comparator): 10 mg Microcrystalline cellulose in orange capsule, Size 0, 2 capsules as a single oral dose
  Interventions: Drug: 20 mg AZD7325; Drug: Placebo

INTERVENTIONS:
Drug: 20 mg AZD7325 — A single 20 mg oral dose of AZD7325
Drug: Placebo — A single oral dose

SUMMARY:
GABA (gamma-aminobutyric acid) is the main inhibitory neurotransmitter in the human brain. For years, drugs that enhance its effects (e.g., benzodiazepines such as diazepam/Valium) have been used to treat various diseases such as epilepsy, insomnia, anxiety or movement disorders. However, the use of these medications is often compromised because of their side effects, such as sleepiness, memory problems, and addiction.

Therefore, effort has been made to develop drugs that act more selectively in the brain to exert the positive therapeutic effects and are devoid of the unwanted side effects. AZD7325 is one of these drugs. It has been tested in more than 700 people and so far proved to be generally well tolerated. Positron emission tomography (PET) study in humans demonstrated that AZD7325 binds to GABA A receptors in the brain after a single dose. Early clinical studies have shown that it has less sedative and cognitive adverse events as compared with a benzodiazepine lorazepam.

The investigators now wish to evaluate if effects of AZD7325 can be objectively measured in healthy volunteers and to establish which of the drug's outcomes could be utilised for further studies in patients with neurological diseases.

The investigators are especially interested in the effects of AZD7325 on manual dexterity and skin sensation of the hand. This can be assessed by a number of simple non-invasive tests of object manipulation and detection of different sensory stimuli such as touch, vibration, or temperature. Recent studies show that healthy individuals who performed better in similar tasks had more GABA in relevant areas of their brain. If performance in these tasks in healthy volunteers can be improved by enhancing GABA effects in the brain with AZD7325, this would create the grounds for the use of this medication to treat symptoms of certain neurological disorders in which motor control and sensation of the hand is impaired (e.g., polyneuropathy).

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged 18 to 55 years (extremes are included)
* A body weight resulting in a body mass index (BMI) of 18-30 kg/m2 (extremes included) using the formula BMI = body-weight [in kg] / body-height [in m]2
* Able and willing to sign the Informed Consent Form prior to screening evaluations.
* History of good physical and mental health as determined by history taking and laboratory examinations, ECG, blood pressure and heart rate recordings as judged by the investigator
* Willing not to consume alcohol or to smoke or chew tobacco on days of assessments
* Subjects must be willing to avoid unprotected vaginal intercourse with women of child bearing potential (see above under 3.5) or donating sperm for the duration of the study and a further 1 week after drug administration.

Exclusion Criteria:

* History of allergy/idiosyncrasy to AZD7325 or chemically related compounds or excipients which may be employed in the study or to any other drug used in the past
* Subject has taken systemically (po, iv) any potent or moderate CYP3A4 or CYP2C9 inhibitor, 1 month prior to screening (topical or inhaled are permitted) such as: aprepitant, barbiturates, carbamazepine, clarithromycin, erythromycin, cyclosporine, diltiazem, efavirenz, fluconazole, HIV protease inhibitors, glucocorticoids, itraconazole (oral/IV), ketoconazole, nefazodone, nevirapine, phenytoin, pioglitazone, primidone, rifabutin, rifampicin, telithromycin, St. John's wort, verapamil
* Use of any prescription drug judged by the investigator as potentially interfering with this trial within two weeks prior to the first dosing, except for topical medication without systemic exposure
* Clinically relevant history or presence of any medical disorder, potentially interfering with this trial
* Clinically relevant abnormal laboratory, ECG, HR or BP at screening as judged by the investigator
* History of or current abuse of drugs (including prescription medication) or alcohol or solvents
* Smoking in excess of 5 cigarettes per day or the equivalent within 28 days prior to the screening visit
* Smoking or chewing of tobacco or consume of alcohol, 24 hours before and on the days of assessment
* Subject is family member or in the employment line management of study personnel
* Subject has abnormal screening laboratory values
* Subject's partner is planning pregnancy within 3 months of last dosing
* Participation in an IMP intervention trial within last month or more than four in the previous 12 months
* Abnormal responses in the object manipulation task and psychophysical measures, SDMT, VAS outside 95% confidence interval of normal at screening visit
* Subjects with a history of epilepsy, seizures or episodes of unexplained and unprovoked loss of consciousness

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in peak grip force in an object manipulation task | from baseline at 1, 2, and 3 hours after the study medication

SECONDARY OUTCOMES:
Changes in parameters of object manipulation in a object manipulation task (grip force rate) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: grip force rate
Changes in parameters of object manipulation in a object manipulation task (load force rate) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: load force rate
Changes in parameters of object manipulation in a object manipulation task (static load force) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: static load force
Changes in parameters of object manipulation in a object manipulation task (static grip force) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: static grip force
Changes in parameters of object manipulation in a object manipulation task (9-hole pegboard test) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: 9-hole pegboard test
Changes in performance in the psychophysical tests of cutaneous sensation ("bumps" test) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: "bumps" test
Changes in performance in the psychophysical tests of cutaneous sensation (grating orientation task) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: grating orientation task
Changes in performance in the psychophysical tests of cutaneous sensation (vibrotactile sensitivity) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: vibrotactile sensitivity
Changes in performance in the psychophysical tests of cutaneous sensation (thermal sensitivity) | from baseline at 1, 2, and 3 hours after the study medication
  Parameters: thermal sensitivity
Change in the rating on a 0-100 mm Visual Analogue Scale (VAS) of degree of sedation | from baseline at 1, 2, and 3 hours after the study medication
Change in the score of Symbol Digit Modalities Test (SDMT) | from baseline at 1, 2, and 3 hours after the study medication
Safety and tolerability of a single dose of AZD7325 by assessment of adverse events, vital signs, physical examination, ECG, and laboratory variables | 3 times during the trial period, an expected average of 4 weeks (before each dose and 48-96 hours after the last dose of study medication). Adverse events also at follow-up telephone call within a week after the last dose of study medication
  Composite outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Koltzenburg, Prof, Principal Investigator — Institute of Neurology, University College London
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom